CLINICAL TRIAL: NCT06482775
Title: Dexmedetomidine for Analgosedation to Newborn Infants During Neonatal Intensive Care - a Prospective Pharmacokinetic/ Pharmacodynamic/ Pharmacogenetic Observational Study.Cohort 3 in The SANNI Project.
Brief Title: Dexmedetomidine for Analgosedation to Newborn Infants During Neonatal Intensive Care
Status: Withdrawn | Type: Observational
Why Stopped: Problems with the study costs after Covid-19
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); Karolinska Institutet (Other); Helsinki University Central Hospital (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); Örebro University, Sweden (Other); The Swedish Research Council (Other Government); University of Tartu (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-002506-37
Record Dates: First submitted 2020-08-04; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2021-06

CONDITIONS: Intensive Care, Neonatal; Analgesia; Hypnotics and Sedatives
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- dexmedetomidine: Infusion of dexmedetomidine 4 microgram/mL.
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: dexmedetomidine — The dosing and administration will be implemented according to an algorithm based on pain scoring results

SUMMARY:
A prospective pharmacokinetic (PK), pharmacodynamic (PD) and pharmacogenetic (PG) observation study, including the PK/PD/PG relationship, on dexmedetomidine administered for analgesia and sedation to postsurgical and other newborn sick infants needing the drug for clinical reasons during neonatal intensive care. Phase III - therapeutic confirmatory study.

DETAILED DESCRIPTION:
The patients will be treated according to clinical guidelines and judgement as decided by the responsible clinical doctor.

The dosing and administration of dexmedetomidine will be implemented according to an algorithm based on pain scoring results.

Apart from extra blood sampling and extended bedside monitoring for amplitude-integrated EEG (aEEG), Near InfraRed Spectroscopy (NIRS), and Galvanic Skin Response (GSR) the care is according to clinical routine.

In total 100 infants will be included.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infants: - born 34+0 gw with a need for dexmedetomidine for analgesic and/or sedative treatment after postnatal surgical correction of congenital malformations and who will be cared for in the PICU (postoperative intensive care unit) and in a some few cases in the NICU (neonatal intensive care unit), or
* with a corresponding age of 37 gw, who are in need for dexmedetomidine according to clinical judgment and cared for in the NICU.
* Existing arterial or venous cannulas/catheters for repeated nontraumatic blood sampling
* Informed and written parental consent obtained before study start.

Exclusion Criteria:

* Infant older than age corresponding to gw 46+0
* Previous treatment with the dexmedetomidine within 72 hours (only for postoperative infants).
* Congenital cardiac malformations requiring surgery on extracorporeal circulation and treatment with hypothermia.
* Ongoing renal replacement treatment
* Any serious medical condition or ethical issues that could, in the investigators opinion, interfere with the study procedures.

Max Age: 27 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Sick newborn infants in need of intensive care.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of dexmedetomidine | Repeated blood samples (5 minutes after the loading dose until 12 hours after stop of infusion)
  The plasma concentration will be analysed and then further reported using NONMEM® (Non-linear Mixed Effect Modelling) population-based PK modelling.
Neurophysiologic response; global brain network function in relation to PK | Baseline until 12 hours after stop of infusion
  Assessment of global brain network function will be based on Activation Synchrony Index.

SECONDARY OUTCOMES:
Change in heart rate, HR, (hemodynamic response) in relation to PK (PK/PD) | Baseline until 12 hours after stop of infusion
  HR will be monitored 1/second according to clinical routine in the neonatal intensive care, and concomitantly downloaded into the aEEG (amplitude integrated electroencephalography) monitor. The change will be described as percentage increase/decrease. The change from baseline response in heart rate using longitudinal models of data on these endpoints following dexmedetomidine administration using a population PK/PD approach.
Change in mean arterial blood pressure, MABP, (hemodynamic response) in relation to PK (PK/PD) | Baseline until 12 hours after stop of infusion
  MABP will be monitored 1/second according to clinical routine in the neonatal intensive care, and concomitantly downloaded into the aEEG (amplitude integrated electroencephalography) monitor. The change will be described as percentage increase/decrease. The change from baseline response in MABP using longitudinal models of data on these endpoints following dexmedetomidine administration using a population PK/PD approach.
Change in/association between Near Infrared spectroscopy, NIRS, in relation to PK. | Once per second (from baseline until 12 hours after stop of infusion)
  NIRS will be monitored 1/second according to clinical routine in the neonatal intensive care, and concomitantly downloaded into the aEEG (amplitude integrated electroencephalography) monitor. The change will be described as percentage increase/decrease
Procedural pain response in relation to PK: assessed with change in galvanic skin response | Once during treatment with dexmedetomidine
  Procedural pain response at a short standardized pain stimulation;

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Norman, MD, Principal Investigator — Region Skane
Locations (2):
- Sweden (2):
  - Skane University Hospital, Lund
  - Karolinska Universitetssjukhuset, Stockholm

IPD SHARING:
Plan to Share IPD: No